CLINICAL TRIAL: NCT04858113
Title: Pilot Project: Comparing the Short-term Effects on the Tear Film and Lid Margin Between Diluted Baby Shampoo and Blephaclean
Brief Title: Short-term Effects on Tear Film (Baby Shampoo vs Blephasol)
Acronym: Blepha
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Dr Daniela Oehring, Dr, University of Plymouth
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SoHP_DO_05
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baby Shampoo (Placebo Comparator): Conventional Baby shampoo
  Interventions: Other: Baby Shampoo
- No intervention (No Intervention): Baseline condition without intervention
- Blephaclean (Experimental): Intervention
  Interventions: Other: Blephaclean

INTERVENTIONS:
Other: Blephaclean — Blephaclean wipes are used to help treat symptoms of blepharitis (eyelid inflammation) which is commonly associated with dry eye disease and meibomian gland dysfunction.
  Arms: Blephaclean
Other: Baby Shampoo — Conventional baby shampoo
  Arms: Baby Shampoo

SUMMARY:
Lid cleansing is the standard regime that is recommended for the management of blepharitis in the UK and beyond. Whilst many successful commercial preparations exist, and some with clinical evidence, professional guidelines (UK Royal College of Ophthalmologists, UK College of Optometrists, AAO, etc.) continue to advocate the use of a diluted solution of baby shampoo, despite no clinical evidence of its safety, tolerance or long term effectiveness, and despite a statement form the manufacturers that it should not be used for this purpose. Where licensed, registered products exist it seems bizarre that we have this situation, but a Cochrane review from 2012 indicated that only a longitudinal, randomized controlled trial against baby shampoo would alter their conclusions. Whilst that sort of clinical study is possible, it is proposed here to start with a short-term study to look at the immediate changes induced in the tear film and ocular surface when comparing baby shampoo with Blephasol solution, in a blind, randomized controlled trial.

DETAILED DESCRIPTION:
Aims/Key Questions: The hypothesis is: Diluted baby shampoo is more disruptive and deleterious to the human tear film and ocular surface than Blephaclean solution. It is expected that there will be a clinically meaningful difference (approximately 30%) in the non-invasive tear-break up time after the application of baby shampoo compared to Blephaclean.

Potential outcomes: To raise awareness that the safety profile of baby shampoo is insufficient to make it a professional and ethical recommendation for daily lid hygiene.

Recruitment: All subjects will be recruited from the staff and student population of the Faculty of Health and Human Sciences, Plymouth University as well as patients of The Centre for Eyecare Excellence (CEE) and Well-being centre (WBC) at Plymouth University. The recruitment will be carried out via email, flyers and direct invitation. After the first contact, the information sheet, as well as the informed contents, will be sent, or a printed version will be given to all potential subjects.

Design: This prospective study is a two-visit, prospective, cross-sectional, double-blinded and randomized controlled trial. The basic population is described as a healthy UK population with diverse ethnic backgrounds and physiological variation. The principal investigator will carry out the data collection at the Peninsula Allied Health Centre, CEE or WBC (Plymouth University). Ethical approval was grantet. This study conforms to the ethical principles of the Declaration of Helsinki, ICH guidelines for Good Clinical Practice (GCP) and Plymouth University's Principles for Research Involving Human Participants.

Sample size calculations were performed for detecting differences between two dependent not-normally distributed means. A maximum effect size (NIK-BUT difference after the application of baby shampoo compared to Blephaclean) of 0.4 is expected with alpha=0.05 and beta=0.20 (80% power). A sample size of 52 will be required. If considering potential dropouts, the study will aim to recruit 60 subjects. The effect size was calculated based on the distribution of the NIK-BUT in healthy eyes (Abdelfattah et al. 2015).

Primary outcome measure: The non-invasive Keratograph (tear film) break-up time (NIK-BUT) is defined as the primary outcome parameter for the present study. The NIKBUT is defined as the interval between the last complete blink and the first appearance of a dry spot, or disruption in the tear film detected automatically by the Keratograph 5M (in seconds).

Randomisation Method: The choice of the eye side, as well as the first cleansing product, will be randomised to minimise investigator bias. Block-wise randomisation is chosen to guarantee an equal group size. The block size is calculated with m = 2n (n means a number of possible groups) per group.

Subject History & Study Eligibility (Fig. 1 - 1 & 2): Before determining study eligibility for each subject, the information sheet and the informed content will be handed out to the patient subject again. During recruitment potential subjects will also be given the information sheet. This will ensure that the participant has had sufficient time to understand the study and make an informed decision about participating in the study. Eligible subjects will be allowed to continue. Non-eligible subjects will be dismissed at this time. Subjects will have procedures performed on both eyes. Testing order was designed to sequentially administer the least invasive test to the most invasive test. This methodology will ensure that a previous procedure will have a minimal effect on all subsequent assessments.

Visual Acuity with height and low contrast: The investigator will measure the subject's visual acuity (VA) on a calibrated LogMAR chart at 100% contrast and FrACT for low contrast VA. If the patient is unable to read the 6/12 letters monocular, the investigator will pinhole over the patient's unaided or presenting refractive error correction to determine the subject's visual potential. After finishing both eyes separately, the visual acuity will be examined binocularly with the same procedure.

Questionnaires: Subjects will be asked to complete the OSDI and McMonnies questionnaires.

Tear film & ocular surface assessment: The tear film will be examined with the Oculus Keratograph 5M from Oculus Optikgeräte GmbH (following K5M). This will include automatic assessments of the Non-Invasive Keratograph Break-Up time (NIKBUT), the tear meniscus height, lipid layer assessment, tear flow and bulbar (conjunctival) redness. Additionally, the K5M will also be used to assess corneal and conjunctiva staining. For assessing bulbar and palpebral conjunctival staining a sterile Lissamine green strip will be wet with sterile saline and applied to the superior bulbar conjunctiva.

Lid cleansing procedure: One investigator will prepare the products such that the principal investigator and the participant are masked. The Principal investigator will apply the product to the upper and lower lid areas and margins, using standard techniques. One eye will be treated using Blephaclean the other eye will be treated using baby shampoo, randomised for visit 1 and visit 2. The Principal investigator needs to apply and gently massage foam from one bottle onto the periocular skin of the closed superior and inferior eyelids of the designated eye with clean fingertips for one minute before rinsing with water, and to take care to avoid the transfer of residual products to the fellow eye during cleansing and drying. The Principal investigator has to avoid direct contact with the ocular surface, and to clean their hands prior to using the second treatment for the fellow eye, in order to prevent cross contamination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be over 18 and under 60 years of age
* Completed a comprehensive eye exam in the last two years
* Contact lens wearers must have stopped wearing for a minimum of two days if wearing soft contact lenses and one week if wearing RGP lenses.
* The subject must have an adequate understanding of the English language to be able to comprehend the oral and written instructions.

Exclusion Criteria:

Determination during enrolment:

* Pregnancy or breast-feeding whilst the examination
* Application of any eye drops within the last 48 hours before the examination
* Application of medication within the last 30 days which influences the body water regulation system (e.g. antidepressants, diuretics, corticosteroids, histamine-receptor antagonist, immune-modulators)
* Change of ocular therapy within the last 30 days before the examination
* Permanent application of eye drops or ocular medication
* On-going ocular treatment
* Any kind of ocular pathology or history of refractive surgery
* Any kind of systemic disease which affect collagen and the body water regulation system (Marfan syndrome, osteogenesis imperfect, pseudoxanthoma elasticum, Ehlers-Danlos, diabetes, rosacea, acne, cardiovascular disease, thyroid disease)

Early termination of the study:

* Drop-out: active termination (decision made by the test person)
* Decision made by the examiner (inadequate compliance, change in the medical condition, as a result, the exclusion criterion is fulfilled)
* Decision made by the lead investigator/ sponsors

It is possible to withdraw the participation in the study at any time. The participant is not liable to give any reasons for withdrawing. If the study is withdrawn because of the decision of the investigator, the reasons must be given in the screening form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
NIKBUT | 1 day
  Non-invasive break up time

CONTACTS AND LOCATIONS:
Locations (1):
- University of Plymouth, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No